CLINICAL TRIAL: NCT06651268
Title: Local Application of Vancomycin (powder) Before Surgical Closure Helps to Reduce Sternal Wound Infection After Cardiac Surgery Procedures.
Brief Title: Effectiveness of Topical Vancomycin in Reducing Sternal Wound Infections Post-Cardiac Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Qaiser Aziz, Head of Cardiac Surgery, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LNH-2024
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-01

CONDITIONS: Wound Complication; Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- while Group B (vancomycin group, n=12) had vancomycin powder applied during closure. T (Experimental)
  Interventions: Drug: while Group B (vancomycin group, n=12) had vancomycin powder applied during closure. T
- : Group A (control, n=12) received standard closure techniques without vancomycin powder (Other): Group A (control, n=12) received standard closure techniques without vancomycin powder
  Interventions: Drug: while Group B (vancomycin group, n=12) had vancomycin powder applied during closure. T

INTERVENTIONS:
Drug: while Group B (vancomycin group, n=12) had vancomycin powder applied during closure. T — while Group B (vancomycin group, n=12) had vancomycin powder applied during closure. T

SUMMARY:
Title: The Role of Vancomycin Powder in Reducing Sternal Wound Infections Following Cardiac Surgery: A Randomized Controlled Trial

Introduction:

Sternal wound infections (SWIs) are significant complications in cardiac surgery, leading to serious issues like mediastinitis, prolonged hospital stays, and higher healthcare costs. This study explores the potential of topical vancomycin powder to reduce SWIs when added to the standard use of systemic antibiotics.

Objectives:

To assess the effectiveness of vancomycin powder in preventing SWIs post-cardiac surgery.

To determine its impact on postoperative hospital stays.

Study Design and Methodology:

A randomized controlled trial will be conducted at Liaquat National Hospital, Karachi, with 24 patients (12 in each group).

Group A will receive standard wound closure, while Group B will receive vancomycin powder applied to the sternal wound.

Postoperative wound assessments will be conducted at 48 hours, 7 days, and 1 month.

Ethical Considerations:

Ethical approval will be obtained, and informed consent will be sought from all participants

DETAILED DESCRIPTION:
The sternotomy approach is widely used in cardiac surgeries, making sternal wound infections a significant concern. These infections can lead to serious complications, including sepsis, reoperation, and increased healthcare costs. Systemic antibiotic prophylaxis is a common practice, but local antibiotic application at the surgical site could further reduce the risk of infection. Vancomycin, due to its effectiveness against gram-positive bacteria, is an ideal candidate for local application. Previous studies in orthopedic surgeries have demonstrated reduced infection rates with vancomycin powder, but its efficacy in cardiac surgery has not been thoroughly explored. This study aims to investigate whether local application of vancomycin powder reduces the incidence of sternal wound infections after cardiac surgery compared to standard care. Additionally, it will evaluate secondary outcomes such as hospital stay duration, postoperative morbidity, and wound-related complications, including dehiscence and the need for reoperation.

The study will be a randomized controlled trial conducted at Liaquat National Hospital, Karachi, Pakistan. A total of 24 patients undergoing cardiac surgery will be randomly allocated to either a control group (standard closure technique) or an intervention group (1 gram of vancomycin powder applied locally before sternal closure). Both groups will receive systemic antibiotic prophylaxis as part of routine care.

This study aims to provide evidence on the efficacy of local vancomycin powder application in reducing sternal wound infections after cardiac surgery. If successful, it could offer a simple, cost-effective intervention to improve postoperative outcomes in cardiac surgery patients. Further research may be needed to validate the findings and support its widespread implementation.

ELIGIBILITY:
Inclusion Criteria:

* .Patients aged between 21 and 80 years were included in the study.
* Both male and female participants were eligible.
* Patients undergoing various adult cardiac surgical procedures, including coronary artery bypass grafting (CABG), atrial septal defect (ASD) repair, ventricular septal defect (VSD) repair, and valve replacement, were considered for inclusion.

Exclusion Criteria:

* Patients who did not provide informed consent were excluded from the study.
* Individuals with a known sensitivity to vancomycin were not eligible.
* Pediatric patients were excluded.
* Patients undergoing redo surgeries were also excluded from participation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of sternal wound infections (SWIs) following cardiac surgery | he patients will be evaluated at three key time points: 48 hours post-surgery 7 days post-surgery 1 month post-surgery
  Incidence of sternal wound infections (SWIs) following cardiac surgery in patients who receive vancomycin powder application compared to those who do not. The infections would be diagnosed based on clinical signs such as redness, pain, swelling, and purulent discharge at the wound site.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac Surgery, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to privacy issue